CLINICAL TRIAL: NCT06538532
Title: Effect of Zamzam Water on Streptococcus Mutans and Oral pH in High Caries-Risk Patients
Brief Title: Anticariogenic Properties of Zamzam Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Reham Youssef, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P-OP-24-01
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Caries,Dental; Caries Active
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (A1) Zamzam water mouthwash (Experimental)
  Interventions: Other: Zamzam water
- (A2) Control group: will be on tooth brushing only (No Intervention)

INTERVENTIONS:
Other: Zamzam water — Zamzam water
  Arms: (A1) Zamzam water mouthwash

SUMMARY:
The present study aims to evaluate and compare the effect of Zamzam water as mouthwashes in high caries-risk patients regarding:

i. Streptococcus mutans (S. mutans) count. ii. Oral pH. After 3 and 6 months interval.

DETAILED DESCRIPTION:
The present study aims to evaluate and compare the effect of Zamzam water mouthwashes in high caries-risk patients regarding:

i. Streptococcus mutans (S. mutans) count. ii. Oral pH. all patients will be into two groups; The first group will use Zamzam water mouthwash for a six months with other preventive protocols including fissure sealants and preventive restorations wherever needed, while the second group will undergo preventive protocols only. During these six months, patients will be reassessed at three and six-month intervals regarding S. mutans count, oral pH, and caries risk level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged between 18-35 years.
* Systemically- free individuals.
* High caries-risk patients according to ADA (American Dental Association).
* Not on a medication interfering with salivary secretion.
* Co-operative patients approved to participate in the study.

Exclusion Criteria:

* Patients who are already on any mouthwash regime.
* Patients who are on any medication that would alter the salivary secretion.
* Allergy to any of the ingredients of the study products.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Streptomutans count | 3 months and 6 months
  measurements of Colony forming unit (CFU) will be performed using blood agar and mitis salivarius-bacitracin agar (MSBA).
Salivary PH level | 3 months and 6 months
  using pH meter
caries risk level | 3 months and 6 months
  According to ADA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental medicine for Girls Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided